CLINICAL TRIAL: NCT01286597
Title: The Effects of Lactose Intolerance on Gastrointestinal Function and Symptoms in a Chinese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Principal Investigator, DAI Ning, Director of Gastroenterology department, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 120100047
Record Dates: First submitted 2011-01-18; First posted 2011-01-31 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Lactose Intolerance; Irritable Bowel Syndrome
Keywords: lactose intolerance; DNA sequencing; psychosocial factors; irritable bowel syndrome; visceral hypersensitivity
MeSH Terms: conditions — Lactose Intolerance; Irritable Bowel Syndrome | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dietary (Experimental)
  Interventions: Dietary Supplement: dietary restriction

INTERVENTIONS:
Dietary Supplement: dietary restriction — restrict intake of lactose
  Other Names: exclusion diet；food restriction；dietary treatment

SUMMARY:
Lactose is a carbohydrate found in milk,and Lactase Deficiency (LD) is a condition in which the small intestine cannot digest this carbohydrate due to absent or insufficient amounts of lactase.Individuals with LD may be intolerant of lactose in the diet and experience abdominal cramps, bloating and diarrhea; however the response is variable.Some tolerate moderate amounts of lactose without adverse effect,whereas others experience severe symptoms in response to even small doses. These problems may be representative of wider issues regarding individual tolerance to diet containing ubiquitous poorly absorbed, fermentable carbohydrates (such as: fructose, fructans)and be relevant to symptom generated in patients with diarrhea predominant irritable bowel syndrome (D-IBS).

This project will investigate the effects of diet,lifestyle stress and psychiatric dietary on the development of functional gastrointestinal symptoms. Lactose will be used to assess tolerance to dietary challenge, a test that is particularly relevant in a Chinese population with a high prevalence of lactase deficiency.

DETAILED DESCRIPTION:
Study #1: Questionnaire study in general Chinese population (n=2000).

Study #2: Physiologic study in patients attending gastroenterology clinic (n=600) including in subgroups assessment of genetic factors,tolerance to lactose challenge and assessment of visceral sensitivity.

Study #3: Assessment of appropriate dosage of lactose hydrogen breath test in a population with high-prevalence of lactase deficiency.

Study #4: Impact of a determined dietary intervention on abdominal symptoms compatible with D-IBS.

study #5: The association of visceral sensitivity induced by LI with mucosal immune activation and psychological factors in D-IBS patients

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 16 years old and not more than 75 years old.
2. Ability to communicate with the investigator, complete study questionnaires (with help of investigator) and provide informed consent.

Exclusion Criteria:

1. Progressive, severe disease requiring active medical management (e.g. advanced cardiac, liver, renal or neurological disease, advanced cancer)
2. History of significant gastrointestinal pathology (other than gastro-oesophageal reflux disease and functional bowel diseases)
3. History of gastro-intestinal surgery (except appendicectomy, cholecystectomy, hernia repair).
4. Evidence of active drug or alcohol abuse

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To assess the effects of lactose intolerance on gastrointestinal function and symptoms | Three years

SECONDARY OUTCOMES:
To measure the intake of dietary lactose in the adult general population and in patients with IBS | three years
To assess genetic factors, tolerance to lactose challenge and visceral sensitivity. | three years
To assess appropriate dosage of lactose hydrogen breath test | two years
To determine the impact of a determined dietary intervention on abdominal symptoms compatible with D-IBS. | three years
To explore the association of visceral sensitivity induced by LI with mucosal immune activation and psychological factors in D-IBS patients | two years

CONTACTS AND LOCATIONS:
Overall Officials: Ning DAI, MD, Study Chair — Sir Run Run Shaw Hospital, College of Medicine, Zhejiang University, China
Locations (1):
- Sir Run Run Shaw Hospital , College of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Chen B, Du L, Zhang Y, Cen M, Luo L, Xu M, Kim JJ, Dai N. Natural History and Outcomes of Individuals With Functional Bowel Disorder: A 9-year Population-Based Longitudinal Study. Clin Transl Gastroenterol. 2024 Jul 1;15(7):e00715. doi: 10.14309/ctg.0000000000000715. PMID 38752653
- [Derived] Yang JF, Fox M, Chu H, Zheng X, Long YQ, Pohl D, Fried M, Dai N. Four-sample lactose hydrogen breath test for diagnosis of lactose malabsorption in irritable bowel syndrome patients with diarrhea. World J Gastroenterol. 2015 Jun 28;21(24):7563-70. doi: 10.3748/wjg.v21.i24.7563. PMID 26140004
- [Derived] Yang J, Fox M, Cong Y, Chu H, Zheng X, Long Y, Fried M, Dai N. Lactose intolerance in irritable bowel syndrome patients with diarrhoea: the roles of anxiety, activation of the innate mucosal immune system and visceral sensitivity. Aliment Pharmacol Ther. 2014 Feb;39(3):302-11. doi: 10.1111/apt.12582. Epub 2013 Dec 5. PMID 24308871
- [Derived] Yang J, Deng Y, Chu H, Cong Y, Zhao J, Pohl D, Misselwitz B, Fried M, Dai N, Fox M. Prevalence and presentation of lactose intolerance and effects on dairy product intake in healthy subjects and patients with irritable bowel syndrome. Clin Gastroenterol Hepatol. 2013 Mar;11(3):262-268.e1. doi: 10.1016/j.cgh.2012.11.034. Epub 2012 Dec 13. PMID 23246646